CLINICAL TRIAL: NCT03643939
Title: RandomizEd Adaptive Trial of High-Flow Nasal Oxygen Cannula Compared to Non-Invasive Ventilation for AcuTE Respiratory Failure
Brief Title: High-Flow Nasal Oxygen Cannula Compared to Non-Invasive Ventilation in Adult Patients With AcuTE Respiratory Failure
Acronym: RENOVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Berry Consultants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RENOVATEmain_2018_08
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Insufficiency; Respiratory Failure
Keywords: respiratory insufficiency; respiratory failure; non-invasive ventilation; high flow nasal cannula; nasal high flow; trans-nasal insufflation; NIV; HFNC
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Cannula; Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Adaptive, non-inferiority randomized, open-label, controled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Catheter (Experimental): The HFNC (AIRVO2 Fisher & Paykel, Auckland, New Zealand) consists of an apparatus that allows adjustable FiO2 from 21 to 100% and delivers flow up to 60 L/ min.
  Interventions: Device: High Flow Nasal Catheter
- Non-invasive positive pressure ventilation (Active Comparator): NIPPV will be performed using the devices available on centers. Both a dedicated NIPPV device or invasive mechanical ventilator with NIPPV mode are accepted. The interface should be a oronasal or full face mask.
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: High Flow Nasal Catheter — HFNC will deliver through AIRVO2. FiO2 from 21 to 100% and heated humidified gas flow up to 60 l / min with temperature of the circuit maintained at 37 degrees.
  Oxygen flow will be offered through a humidified nasal catheter. Flow and FiO2 will be titrated according to the protocol to maximize patient´s comfort and SpO2.
  Other Names: Optiflow; Airvo; trans-nasal insufflation; Nasal High Flow; High Flow Nasal Cannula; nasal cannula with high-flow oxygen
  Arms: High Flow Nasal Catheter
Device: Noninvasive ventilation — NIPPV will be performed using a facial mask (either oronasal or full face). NIPPV will deliver pressures and FiO2 tailored to specific ARF subgroups, according to the protocol. Adjustments of the inspiratory pressure (IPAP) and expiratory pressure (EPAP) and FiO2 according to protocol
  Other Names: BiPAP; Non-invasive ventilation; Noninvasive positive pressure ventilation
  Arms: Non-invasive positive pressure ventilation

SUMMARY:
RENOVATE study aims to investigate if the respiratory support device called High-Flow Nasal Oxygen Cannula (HFNC) acts similarly (non-inferior) to another respiratory support device called Non-Invasive positive-pressure Ventilation (NIPPV) in preventing endotracheal intubation in adult patients with Acute Respiratory Failure (ARF) from different causes. HFNC is a somewhat new method of respiratory support in adults that has been used in neonatal ARF for some years. The reason this study is necessary is that, even though NIPPV has been demonstrated to prevent endotracheal intubation (and its associated complications) in a broad range of ARF patients, HFNC has been proposed to have the same beneficial effect of NIPPV while being easier tolerated, allowing patients to talk, eat and drink through mouth while on HFNC. RENOVATE will recruit between 800 to 2000 patients (adaptive design) with different types of ARF in Brazil. Patients will be randomized to HFNC or NIPPV and the rate of endotracheal intubation will be compared between groups as well as other parameters such as vital status and other health care related complications.

[IMPORTANT NOTE] On April 13, 2021, on the first interim analysis, the DSMB recommended the interruption of the immunocompromised hypoxemic ARF subgroup.

DETAILED DESCRIPTION:
RENOVATE will investigate if High-Flow Nasal Oxygen Cannula (HFNC) is non-inferior to Non-Invasive positive-pressure Ventilation (NIPPV) in preventing endotracheal intubation or death in adult patients with Acute Respiratory Failure (ARF) from different causes in 7 days. HFNC is a somewhat new method of respiratory support in adults that has been used in neonatal ARF for some years. Even though NIPPV has been demonstrated to prevent endotracheal intubation (and its associated complications) in a broad range of ARF patients, HFNC may have beneficial effect over NIPPV because it is easier to be tolerated, allowing patients to talk, eat and drink through mouth while on therapy. RENOVATE will recruit between 800 to 2000 patients (adaptive design) with different types of ARF in Brazil. The main hypothesis is that HFNC is non inferior to NIPPV in reducing intubation rate or death within 7 days. However, as an adaptive study, this non inferiority hypothesis may change to superiority if gathered data during the study is promissing in the interim analysis. Therefore, sample size may increase to 2000 participants. Patients will be randomized to HFNC or NIPPV and the rate of endotracheal intubation will be compared between groups as well as other parameters such as vital status and other health care related complications.

[IMPORTANT NOTE] On April 13, 2021, on the first interim analysis, the DSMB recommended the interruption of the immunocompromised hypoxemic ARF subgroup.

Trial Update:

We have collected Covid 19 information since march 2020 as an added question in the CRF. There are two questions: one in the elegibility criteria form asking if Covid 19 is suspected and another one in the discharge form asking if Covid 19 was laboratory confirmed. Since then, there were considerably change in prevalence of acute respiratory failure subgroups since the beginning of the trial in 2019. Covid 19, nowdays, is responsible for 63% of our sample size, followed by hypoxemic non immunocompromised subgroup with 19%, acute pulmonary edema and hypoxemic immunocompromised with 8% and finally COPD with 2%. These prevalences are completely different from our previous assumptions in 2019 trial simulations as published in our protocol and statistical analysis plan in March 2022 Volume 24 Number 1 at Critical Care Resuscitation journal. Therefore, the Steering Committee decided that all Covid 19 patients, independent of previous subgroup allocation, would be analysed separately in a 5th subgroup. Update in simulations with different scenarios and new statistical models were done by March 13th 2023 to account for the 5th interim analysis which you can access in the document section of ClinicalTrials.gov. No change in inclusion criteria were made. The only change was the introduction of those two questions described before. These updates are aimed at accommodating the presence of COVID-19 patients in the trial as the main subgroup of patients.

ELIGIBILITY:
[IMPORTANT NOTE] On April 13th 2021, in the first interim analysis, the DSMB recommended for the interruption of the subgroup Immunocompromised De Novo Hypoxemic ARF due to futility.

Sequential adult patients 18 years of age or older admitted to the ICU or emergency department with acute onset respiratory distress suspected of having De Novo hypoxemic ARF (non-immunocompromised) , Immunocompromised De Novo hypoxemic ARF, COPD ARF, Cardiogenic acute pulmonary edema (APE).

Inclusion criteria for these 4 ARF subgroups are detailed below:

A. Inclusion Criteria for Non-Immunocompromised De Novo Hypoxemic ARF.

Patients must meet criteria 1, 2 and 3:

1. Hypoxemia evidenced by SpO2 <90% or PaO2 <60 mmHg in room air
2. Use of accessory muscles, paradoxical breathing, and/or thoracoabdominal asynchrony
3. RR> 25 per minute

B. Inclusion Criteria for Immunocompromised De Novo Hypoxemic ARF.

Patients must meet criteria 1, 2, 3 and 4:

1. Immunosuppression diagnosis:

   i. Use of Immunosuppressive drug or long-term [>3 months] or high-dose [>0.5 mg/kg/day] steroids ii. Solid organ transplantation iii. Extensive solid tumor or solid tumor requiring chemotherapy in the last 5 years iv. Hematological malignancy regardless of time since diagnosis and received treatments v. HIV infection vi. Primary immunodefiency
2. Hypoxemia evidenced by SpO2 <90% or PaO2 <60 mmHg in room air
3. Use of accessory muscles, paradoxical breathing, and/or thoracoabdominal asynchrony
4. RR> 25 per minute

C. Inclusion Criteria for COPD exacerbation:

Patients must meet criteria 1 or 2 and 3 and 4:

1. Previous Diagnosis of COPD based on GOLD guidelines
2. Strong clinical suspicion of COPD i. Smoker or ex-smoker or other CPOD related exposure ii. Presence of chronic dyspnea on exertion or chronic productive cough iii. Excluded other causes for the chronic symptoms (ex. pulmonary fibrosis, heart failure)
3. RR> 25 per minute or use of accessory muscles, paradoxical breathing, and/or thoracoabdominal asynchrony
4. ABG analysis with pH < 7,35 , paCO2> 45 mmHg

D. Inclusion Criteria for ARF secondary to Cardiogenic APE.

Patients must meet criteria numbers 1, 2 and 3:

1. Diagnosis of Cardiogenic Acute Pulmonary Edema (Nava, 2003):

   i. Dyspnea of sudden onset ii. Widespread rales with or without third heart sound 1 iii. Absent history of pulmonary aspiration, infection or previous history of pulmonary fibrosis iv. Pulmonary edema as the main clinical hypothesis v. Previous heart failure clinical history or acute coronary syndrome vi. If chest X-ray is already available at randomization, it must be suggestive of bilateral pulmonary edema
2. RR > 25 per minute
3. SpO2 < 95%

Exclusion Criteria for all subgroups of ARF

1. Indication of emergency ETI:

   * Prolonged respiratory pauses
   * Cardiorespiratory arrest
   * Glasgow ≤12
   * HR < 50 bpm with decreased level of consciousness
   * pH < 7.15 irrespective of the cause
2. Psychomotor agitation that prevents adequate medical / nursing care requiring heavy sedation
3. Persistent hemodynamic instability with MAP <65 mmHg, SBP <90 mmHg after adequate volume resuscitation or requiring norepinephrine> 0.3 microg / kg / min or equivalent.
4. Contraindications to non-invasive ventilation: face deformities or traumas, recent esophageal surgery, hypersecretion, vomiting with aspiration risk
5. Presence of pneumothorax or extensive pleural effusion
6. Severe arrhythmias at risk of hemodynamic instability
7. Thoracic trauma understood as the main cause of ARF
8. Asthma attack
9. Pregnancy
10. Cardiogenic Shock
11. Acute Coronary Syndromes with plans to undergo coronary angiography within 24 hs
12. ARF after orotracheal extubation (up to 72 hours after extubation)
13. Post-surgical ARF (surgery within 72 hours)
14. Hypercapnic ARF due to neuromuscular disease or chest deformities
15. Patients on exclusive palliative care
16. Do Not Intubate order (DNI)
17. Chronic pulmonary disease except COPD
18. Use of more than 6 hours of NIPPV before randomization if hypoxemic ARF in the non-immunosuppressed, in the immunosuppressed hypoxemic, or if exacerbated COPD
19. Use of NIPPV before randomization in the cardiogenic acute pulmonary edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1801 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Endotracheal intubation rate or death | in 7 days
  proportion of endotracheal intubation or death

SECONDARY OUTCOMES:
Mortality | in 28 days
  Death
Mortality | in 90 days
  Death
ICU free days | in 28 days
  Days out of ICU
IMV free days | in 28 days
  Days without IMV inside of ICU after 48 hours of being extubated

OTHER OUTCOMES:
Length of hospital stay | in 90 days
  Time in hospital in days
Length of ICU stay | in 90 days
  Time in the ICU in days
Vasopressor free days | in 28 days
  Days without use of vasopressor inside of ICU
Proportion of patients who received do-not-intubate-order | in 7 days
  Proportion of patients that received DNI order after randomization was done
Patient confort score | 7 days
  Visual scale varying from 0 (no disconfort) to 100 (maximal disconfort)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, MD, Study Chair — Research Institute - Hospital do Coracao, Sao Paulo, Brazil; Israel Maia, MD, Principal Investigator — Research Institute - Hospital do Coracao, Sao Paulo, Brazil; Leticia Kawano-Dourado, MD, Principal Investigator — Research Institute - Hospital do Coracao, Sao Paulo, Brazil; Laurent Brochard, MD, Study Chair — St. Michael's Hospital (Toronto, Canada); Carlos R Carvalho, MD, Study Chair — Pulmonary Division University of Sao Paulo, Sao Paulo, Brazil
Locations (1):
- Hospital do Coracao, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] RENOVATE Investigators and the BRICNet Authors; Maia IS, Kawano-Dourado L, Tramujas L, de Oliveira NE, Souza RN, Signorini DF, Pincelli MP, Zandonai CL, Blasius RT, Freires F, Ferreira VM, Romano MLP, Miura MC, de Censo CM, Caser EB, Silva B, Santos Bonomo DC, Arraes JA, de Alencar Filho MS, Alvares Horta JG, Oliveira DC, Boschi E, Costa RL, Westphal GA, Ramos J, Lacerda FH, Filho CRH, Pinheiro BV, de Andrade Neumamm LB, Guimaraes Junior MRR, de Souza DT, Ferreira JC, Ohe LN, Schettini DA, Thompson MM, de Oliveira MCF, Veiga VC, Negrelli KL, Santos RHN, Damiani L, Gurgel RM, Gomes SPC, Lima LM, Miranda TA, Laranjeira LN, de Barros E Silva PGM, Machado FR, Fitzgerald M, Bosse A, Marion J, Carvalho CRR, Brochard L, Lewis RJ, Biasi Cavalcanti A. High-Flow Nasal Oxygen vs Noninvasive Ventilation in Patients With Acute Respiratory Failure: The RENOVATE Randomized Clinical Trial. JAMA. 2025 Mar 11;333(10):875-890. doi: 10.1001/jama.2024.26244. PMID 39657981
- [Derived] Maia IS, Kawano-Dourado L, Zampieri FG, Damiani LP, Nakagawa RH, Gurgel RM, Negrelli K, Gomes SPC, Paisani D, Lima LM, Santucci EV, Valeis N, Laranjeira LN, Lewis R, Fitzgerald M, Carvalho CRR, Brochard L, Cavalcanti AB; RENOVATE Investigators and the BRICNet. High flow nasal catheter therapy versus non-invasive positive pressure ventilation in acute respiratory failure (RENOVATE trial): protocol and statistical analysis plan. Crit Care Resusc. 2023 Oct 18;24(1):61-70. doi: 10.51893/2022.1.OA8. eCollection 2022 Mar 7. PMID 38046839

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03643939/SAP_000.pdf